CLINICAL TRIAL: NCT06576648
Title: Optimizing Mobile Interventions to Overcome Stigma and Promote HIV Prevention
Brief Title: Thailand HIV and Stigma Reduction Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Principal Investigator, Bo Wang, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001982; R34MH134682-01A1 (NIH)
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: Pre-Exposure Prophylaxis; HIV Prevention; mHealth; Stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard PrEP counseling, mHC, and FRESH content (Experimental): Participants in this arm will receive standard PrEP counseling, followed by four mHC sessions and six FRESH sessions to reduce stigma and increase utilization of HIV prevention services.
  Interventions: Behavioral: Mobile Healthy Choices (mHC); Behavioral: Finding Respect and Ending Stigma around HIV (FRESH); Behavioral: Standard PrEP Counseling
- Standard PrEP counseling and mHC (Experimental): Participants in this arm will receive standard PrEP counseling, followed by four mHC sessions to reduce stigma and increase utilization of HIV prevention services.
  Interventions: Behavioral: Mobile Healthy Choices (mHC); Behavioral: Standard PrEP Counseling
- Standard PrEP counseling and FRESH content (Experimental): Participants in this arm will receive standard PrEP counseling, followed by six FRESH sessions to reduce stigma and increase utilization of HIV prevention services.
  Interventions: Behavioral: Finding Respect and Ending Stigma around HIV (FRESH); Behavioral: Standard PrEP Counseling
- Standard PrEP counseling (Experimental): Participants in this arm will receive the standard PrEP counseling.
  Interventions: Behavioral: Standard PrEP Counseling

INTERVENTIONS:
Behavioral: Mobile Healthy Choices (mHC) — mHC is a four-session, 20-minute, motivational interviewing-based intervention, which will be delivered on the CIAS platform. It will be tailored to participants' responses given during the interaction in the intervention. In the first two sessions, the (virtual) counselor will motivate participants to overcome stigma and utilize HIV prevention services by using tailored motivational interviewing strategies, develop an individualized change goal based on their readiness, and provide cognitive behavioral strategies. In the last two sessions, the counselor will review the change plan, monitor progress, and provide support for sustained behavioral change. The sessions will occur within three months after baseline.
  Arms: Standard PrEP counseling and mHC; Standard PrEP counseling, mHC, and FRESH content
Behavioral: Finding Respect and Ending Stigma around HIV (FRESH) — FRESH content includes six 10-15 minute sessions with interactive, culturally sensitive multimedia modules, which will be delivered on the CIAS platform. The content will aim to improve self-efficacy, reduce intersectional stigmas and promote HIV preventative behaviors. The sessions will occur within three months after baseline.
  Arms: Standard PrEP counseling and FRESH content; Standard PrEP counseling, mHC, and FRESH content
Behavioral: Standard PrEP Counseling — All participants will receive one-on-one, face to face counseling from focusing on sexual and behavioral risk assessment for HIV/STIs, risk reduction, and HIV prevention. For those not on PrEP, the sessions will focus on risk perception, awareness of PrEP, and facilitators and barriers to PrEP access. For those on PrEP, the sessions will focus on adherence. The counseling will be provided at baseline, 3 months, and 6 months.

SUMMARY:
This project will develop a multi-component, technology-delivered intervention designed to reduce HIV and intersectional stigma and improve the use of HIV pre-exposure prophylaxis (PrEP) among HIV-negative Thai vulnerable emerging adults (18-29 years).

ELIGIBILITY:
Aim 1 (Formative Research and Beta-Testing) Transgender women

Inclusion Criteria:

* Ages between 18 and 29 years
* Male sex at birth
* Self-identifies as women, transgender women or culturally identifies with the female spectrum
* Laboratory-confirmed HIV-negative status
* Self-reported recent history of condomless sex
* Able to understand, read and speak Thai
* Either not started PrEP or currently on PrEP but not adherent (taking ≤3 pills/week) in the past month.

Exclusion Criteria:

* Have a serious cognitive or psychiatric problem compromising ability to provide informed consent
* Have active suicidal ideation or major mental illness at the time of interview (these patients will be referred for treatment)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g., decreased creatinine clearance)
* Currently enrolled in another HIV intervention study.

Healthcare providers Inclusion criteria

* Age 18 or above
* Has provided HIV prevention or treatment services for TGW for at least one year Exclusion criteria
* None

Aim 2 (Pilot RCT) Transgender women Inclusion criteria

* Ages between 18 and 29 years
* Male sex at birth
* Self-identifies as women, transgender women or culturally identifies with the female spectrum
* Laboratory-confirmed HIV-negative status
* Self-reported recent history of condomless sex
* Able to understand, read and speak Thai
* Either not started PrEP or currently on PrEP but not adherent (taking ≤3 pills/week) in the past month.

Exclusion criteria

* Have a serious cognitive or psychiatric problem compromising ability to provide informed consent
* Have active suicidal ideation or major mental illness at the time of interview (these patients will be referred for treatment)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g., decreased creatinine clearance)
* Currently enrolled in another HIV intervention study.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender women
Enrollment: 154 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability: System Usability Score (SUS) | Month 3, Month 6
  The SUS is a 10-item, 5-point Likert scale for evaluating subjective usability. Each item is scored from 1 to 5, with the calculation involving either subtracting 1 from the user response or the user response from 5 depending on the item. The scores are then summed and multiplied by 2.5 to obtain a total score ranging from 0 to 100. A score above 80 indicates that the intervention is acceptable.
Intervention Acceptability: Exit Interview | Month 3
  Participants will be asked about their experiences using mHC and FRESH content and potential improvements.
Intervention Feasibility: Participant retention | Baseline through Month 6
  Participant retention rate of over 85% at 6-month follow-up will be the minimum criterion for feasibility.
Intervention Feasibility: Number of FRESH sessions viewed | Baseline through Month 6
  Intervention feasibility will be evaluated by the total number of FRESH sessions viewed.
Intervention Feasibility: Number of mHC sessions completed | Baseline through Month 6
  Intervention feasibility will be evaluated by the number of completed intervention sessions.
PrEP Uptake: Self-report | Month 3, Month 6
  PrEP uptake will be assessed using a self-report measure and confirmed via chart review and pharmacy records.
PrEP Adherence: Visual analog scale | Baseline, Month 3, and Month 6
  PrEP adherence will be assessed through the Young Adult Adherence Interview, which contains a visual analog scale (VAS) ranging from 0 to 100. Higher percentages on the VAS indicate greater adherence to ART.
PrEP Adherence: Self-Reported Adherence | Baseline, Month 3, and Month 6
  PrEP adherence will be evaluated through self-reported adherence over the past four weeks. Participants will rate their adherence on a scale ranging from 0 to 100%, with higher percentages indicating better adherence to PrEP. The result will be triangulated with DBS reports.
PrEP Adherence: DBS testing | Baseline, Month 3, and Month 6
  PrEP adherence will be evaluated by tenofovir concentrations in dried blood spots (DBS). The result will be triangulated with self-reports.
HIV testing uptake: Self-report | Baseline, Month 3, and Month 6
  HIV testing uptake will be assessed via self-report and confirmed through chart review.
Intersectional stigma | Baseline, Month 3, and Month 6
  Intersectional stigma will be assessed using the Intersectional Discrimination Index, which includes three subsets: anticipated, day-to-day, and major discrimination. The anticipated and day-to-day discrimination measures each consist of 9 items, while the major discrimination measure includes 13 items. The anticipated discrimination score is calculated as a mean ranging from 0 to 4. The day-to-day discrimination score is based on frequency and can range from 0-9 (lifetime) or 0-18 (past-year). The major discrimination score is based on frequency and can range from 0-26 (lifetime) or 0-13 (past-year). For all three measures, higher scores indicate a greater level of anticipated discrimination or experienced discrimination.
Internalized stigma | Baseline, Month 3, and Month 6
  Internalized stigma will be evaluated using the Internalized AIDS-related Stigma Scale, a 6-item scale. Scores range from 0 to 6, with higher scores indicating greater internalized stigma.
Perceived stigma | Baseline, Month 3, and Month 6
  Perceived stigma will be evaluated using a 13-item, 4-point Likert scale, with a maximum score of 52. Higher scores indicate a higher level of perceived stigma.
Anticipated stigma | Baseline, Month 3, and Month 6
  Anticipated stigma will be evaluated from three different sources (friends and family, neighbors, and others in the community, and healthcare workers) using a 9-item, 5-Likert scale. Scores can reach up to 45, with higher scores indicating a greater expectation of experiencing stigma in the future.
Enacted stigma | Baseline, Month 3, and Month 6
  Enacted stigma will be evaluated with an 8-item, 4-point Likert scale enacted stigma scale. The total score can reach up to 32, with higher scores indicating having more stigma experiences.
PrEP stigma | Baseline, Month 3, and Month 6
  PrEP stigma will be evaluated with a 10-item, 5-point Likert scale. Higher scores indicate a higher level of perceived stigma surrounding PrEP.

SECONDARY OUTCOMES:
Empowerment | Baseline, Month 3, and Month 6
  Empowerment will be assessed using the Healthcare Empowerment Inventory. It's an 8-item, 5-point Likert scale, with total scores ranging from 8 to 40. Higher scores indicate a greater sense of empowerment in her health care.
Information: HIV Knowledge | Baseline, Month 3, and Month 6
  HIV transmission risk awareness will be assessed through an 18-item HIV Knowledge Questionnaire. The total scores can range from 0 to 18, with higher scores indicating a higher level of HIV knowledge.
Information: PrEP Knowledge | Baseline, Month 3, and Month 6
  PrEP knowledge will be assessed through a 13-item PrEP Knowledge Scale. The total score can range from 0 to 13, with higher scores indicating a higher level of PrEP knowledge.
Motivation: Rollnick's Readiness Ruler | Baseline, Month 3, and Month 6
  Motivation will be evaluated using the 5-item Rollnick's Readiness Ruler. Each item ranges from 0 to 10, with higher scores indicating a greater readiness for change in HIV prevention and risk behaviors.
Motivation: Decisional Balance for Problem Behavior | Baseline, Month 3, and Month 6
  Motivation will be assessed using the Decisional Balance for Problem Behavior scale. This 36-item, 5-point Likert scale evaluates the perceived pros and cons of using PrEP.
Behavioral Skills | Baseline, Month 3, and Month 6
  Behavioral skills will be assessed using an adapted version of the Self-Efficacy for Health Promotion and Risk Reduction Questionnaire. This 8-item, 5-point Likert scale measures confidence levels in HIV prevention behaviors, including condom use and adherence to the PrEP schedule. Higher scores indicate a greater confidence in health promotion and HIV prevention.
HIV | Baseline, Month 3, and Month 6
  Fourth-generation HIV-1/2 antigen/antibody combi testing will be used to detect HIV infection.
STI | Baseline and Month 6
  Treponemal test with rapid plasma reagin (RPR) will be used for syphilis, while urine, oropharyngeal, and rectal swabs will be used for gonorrhea and chlamydia.
Sexual Risk | Baseline, Month 3, and Month 6
  Sexual risk will be assessed using a Timeline Followback interview via CASI for any risky sexual behavior over the past 30 days.
Adaptive coping | Baseline, Month 3, and Month 6
  Adaptive coping will be assessed by the Brief Resilient Coping Scale, a four-item, 5-point Likert scale questionnaire. Higher scores indicate greater resilient coping.
Resilience | Baseline, Month 3, and Month 6
  Resilience will be assessed by the Connor-Davidson Resilience Scale. It is a 10-item, 5-point Likert scale questionnaire, with scores ranging from 0 to 40. Higher scores indicate a greater ability to cope with challenges.
Substance use: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Baseline, Month 3, and Month 6
  Substance use will be assessed with ASSIST, an 8-item questionnaire that measures the use of ten substances, including alcohol, smoking, cannabis, and other drugs. Each item is scored from 0 to 12, resulting in a risk score for each ranging from 0 to 31 for tobacco and 0 to 39 for alcohol and other drugs. Higher scores indicate a higher risk of substance use disorder.
Substance use: Alcohol Use Disorder Identification Text (AUDIT-C) | Baseline, Month 3, and Month 6
  Substance use, specifically alcohol use disorder, will be assessed by using AUDIT-C. Each item is scored from 0 to 4, with 0 indicating no alcohol consumption and 4 indicating more hazardous drinking habits. The total score can range up to 12, with higher scores suggesting greater risks of hazardous alcohol consumption.
Mental health | Baseline, Month 3, and Month 6
  Mental health will be evaluated using the Thai General Health Questionnaire. The questionnaire has 12 4-point Likert scale items that assess psychological distress, including depression and anxiety. Scores range up to 48, with higher scores indicating a higher level of psychological distress.
Perceived HIV risk | Baseline, Month 3, and Month 6
  Perceived HIV risk will be assessed using the Perceived Risk of HIV Scale (8 item, 4-point Likert scale). The score ranges up to 40-, with higher scores indicating a high level of perception in HIV risk.
Social support | Baseline, Month 3, and Month 6
  Social support will be assessed using the Social Provision Scale (13-item, 5-point Likert scale). The survey assesses the availability of five forms of social supportsd: attachment, guidance, social integration, reliable alliance, and reassurance of worth. Scores range from 13 to 65, with higher scores indicating receiving a higher level of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (3):
- Thailand (3):
  - Institute of HIV Research and Innovation, Bangkok
  - Rainbow Sky Association of Thailand, Bangkok
  - SWING Foundation, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.